CLINICAL TRIAL: NCT06101836
Title: The Impact of a Short Training Course Focussed on the Acquisition of Conscious Competence on Nurse, Endoscopist and Patient Reported Comfort Scores During and After Colonoscopy
Brief Title: The Impact of Remote Training on Colonoscopy KPIs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BC-07318 E01
Record Dates: First submitted 2023-07-10; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Training; Colonoscopy; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional arm (Other): All participant trainees will undergo the educational intervention, therefore there is only one arm since all participants will undergo the intervention. The intervention is a day where participants (the trainees) will undergo a full day of training in colonoscopy. Comparison of key performance measures in colonoscopy is made before and after the intervention.
  Interventions: Other: Training intervention

INTERVENTIONS:
Other: Training intervention — Trainees underwent a one-day training course (intervention) by consciously competent endoscopists who were physically remote consisting of interactive theoretical sessions and live sessions, where trainees performed colonoscopy in their local endoscopy unit receiving real-time instructions via a tele-conference monitor. Trainers and trainees not doing the colonoscopy, followed the procedure in real-time. KPIs were assessed on trainee-performed colonoscopies for 3 weeks prior and 4 weeks after the intervention.

SUMMARY:
Colonoscopy is a complex, highly operator dependent, practical skill. The consistent attainment of key performance indicators (KPIs) by endoscopists depends primarily upon training. Local factors can make training unstructured and contingent upon the observed practice of a small number of trainers. The investigators sought to demonstrate the feasibility and impact of a virtual-live one day colonoscopy-training course.

DETAILED DESCRIPTION:
The investigators aim to conduct a prospective interventional single-center (University Hospital of Ghent, Belgium) study with trainees to evaluate their colonoscopy associated key performance indicators (KPIs)(Caecum intubation rate, adenoma detection rate, withdrawal time, serious complication rate and patient comfort score) between October and December 2020, prior and post a one-day virtual-live hybrid endoscopy training course.

Trainees and patients have to give their explicit consent for data acquisition and publication.

Consecutive patients undergoing a colonoscopy during the reported period who consent for the study can be included. Colonoscopies are performed with either high-definition or standard-definition white-light colonoscopes. Patients are prepared taking split dose of a polyethylene glycol solution (twice ½ liter) with 2 liters of additional water. During the procedure, patients are consciously sedated (midazolam and fentanyl). All patients receive standard of care endoscopic procedures and therapy.

After each colonoscopy, patients will be asked to fill a questionnaire regarding their comfort during the colonoscopy, using the Global Visual Analog Scale (VAS). Assisting nurses will be asked to note the patient's Gloucester Comfort Score (GCS), a validated comfort score for lower endoscopy. GCS>3 was defined as significant discomfort of the patient. The endoscopist-assessed GCS, and other KPIs of colonoscopy will be extracted from the colonoscopy report. Inclusion of patients starts 3 weeks prior to the planned endoscopy training intervention and continues for another 4 weeks thereafter. Online surveys will be sent to the trainees and trainers after the course, requesting their feedback.

The intervention: a one-day (8 hour) colonoscopy course in the trainees' local (Ghent, Belgium) endoscopy unit, involving virtual-live training by remote (Cheltenham, UK) experts trainers, renowned as consciously competent in colonoscopy technique. Sessions will be a mixture of didactic instruction, interactive discussion and live cases. Every included trainee will perform a live colonoscopy where they are accompanied by a local consultant who acts as a liaison for safety purposes. Live training is delivered via a second television-monitor positioned next to the endoscopic image via teleconference call (Zoom, San Jose, USA). The trainers have access to the real-time image of the endoscopy, as well as the magnetic endoscope imager (scope guide - Olympus, Tokyo Japan). The entire procedure will be recorded allowing the non-participating trainees to follow the course live on their computer. The course will also be available via live-stream (Vimeo, city, USA) external participants, and later for catch-up on the educational endoscopy platform GIEQs.com.

ELIGIBILITY:
Inclusion Criteria:

* trainees: trainees in endoscopy who work at the University Hospital of Ghent who want to participate and who consent for the study
* patients: all patients presenting for a colonoscopy between October and December 2020 and who consent to participate

Exclusion Criteria:

* trainees: trainees in endoscopy who work at the University Hospital of Ghent who do not want to participate and who don't consent for the study
* patients: all patients presenting for a colonoscopy between October and December 2020 and who do not consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Caecum Intubation rate | 3 months
  Trend in measurable colonoscopy key performance indicators pre- and post intervention. Is there a favourable trend in key performance indicator: caecum intubation (intubated YES or No) after the training intervention
Colonoscopy withdrawal time | 3 months
  Trend in measurable colonoscopy key performance indicators pre- and post intervention. What is the withdrawal time (in minutes)? Is there a favourable trend in key performance indicator: colonoscopy withdrawal time (in minutes) after the training intervention
Patient comfort during colonoscopy - Visual analogue scale | 3 months
  Trend in measurable colonoscopy key performance indicators pre- and post intervention. Is there a favourable trend in key performance indicator: patient comfort (Visual analogue scale-number between 0-10, with 0=no pain and 10=worse pain possible) after the training intervention
Patient comfort during colonoscopy - Sedation | 3 months
  Trend in measurable colonoscopy key performance indicators pre- and post intervention. Is there a favourable trend in key performance indicator: patient comfort (amount of sedation necessary/used: midazolam (mg) and/or fentanyl (micrograms)) after the training intervention

CONTACTS AND LOCATIONS:
Overall Officials: David J Tate, Dr., Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital of Ghent, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No